CLINICAL TRIAL: NCT04312763
Title: A Validation of the Functional Low-Vision Observer Rated Assessment (FLORA-20) for Profoundly Blind Individuals
Acronym: FLORA-20
Status: Suspended | Type: Observational
Why Stopped: Study was suspended 4/16/2020 due to global pandemic. Plans to restart or permanently end the study are still being evaluated.
Sponsor: Second Sight Medical Products (Industry)
Collaborators: Boston Biomedical Associates (Other)
Responsible Party: Sponsor
Other Study IDs: CP-11
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Blindness, Acquired
Keywords: Observer-rated instrument
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to validate an observer-rated assessment titled "Functional Low-Vision Observer Rated Assessment (FLORA-20)", which comprises 20 functional vision tasks commonly performed in or around a blind individual's home environment. This study shall be carried out with individuals who have an implanted visual prosthesis device. There are no new implantations or changes to the original implant or external wearables being studied or tested. Additionally, data from the study shall not be used alter standard of care or the user's treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Subjects implanted with the Argus II or Orion device
* Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
* Subject is able to follow instructions and comply with FLORA-20 scheduling and completion of tasks
* Subject is willing to be filmed while performing the FLORA-20 tasks during the study

Exclusion Criteria:

* Subject is unsuitable for study participation as determined by Investigator's clinical judgment (with Sponsor's final input).

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 30 users with the Argus II or Orion system from the US will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2024-12-08 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Inter-observer reliability | Single 1 day visit
  Intraclass correlation coefficient (ICC) of the overall FLORA-20 scores provided by each of the assessors (in-person and remote)
Intra-observer reliability | Single 1 day visit
  ICC of the overall FLORA-20 scores provided by the same assessor, assessed and re-assessed at two different time points

SECONDARY OUTCOMES:
Improvement in Average Performance, ON vs. OFF | Single 1 day visit
  Paired t-test to determine if there is a statistically significant improvement in average performance from ON vs. OFF
Clinical Meaningfulness (Effect Size) | Single 1 day visit
  Cohen's d calculation of overall FLORA-20 scores between device ON vs. OFF
Internal consistency - Cronbach's alpha | Single 1 day visit
  Cronbach's alpha of the individual FLORA-20 task scores
Internal consistency - item-total correlations | Single 1 day visit
  Item-total correlations for each FLORA-20 task

CONTACTS AND LOCATIONS:
Overall Officials: Uday Patel, PhD, Principal Investigator — Second Sight Medical Products, Inc.
Locations (1):
- Second Sight Medical Products, Inc., Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No